CLINICAL TRIAL: NCT04750122
Title: Neoadjuvant Therapy Study Guided by Drug Screening in Vitro Patient-derived Tumor-like Cell Clusters for HER2 Positive Early Breast Cancer Patients
Brief Title: Neoadjuvant Therapy Study Guided by Drug Screening in Vitro for HER2 Positive Early Breast Cancer Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PekingUPH10B003
Record Dates: First submitted 2021-01-26; First posted 2021-02-11 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: HER2-positive Early Breast Cancer
MeSH Terms: interventions — Docetaxel; Trastuzumab; pertuzumab; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoadjuvant therapy base on PTC drug screenning (Experimental): Patients will receive neoadjuvant therapy including trastuzumab, pertuzumab, and chemotherapy based on PTC drug screening.
  Interventions: Drug: neoadjuvant chemotherapy upon in vitro PTC drug sensitivity screenning

INTERVENTIONS:
Drug: neoadjuvant chemotherapy upon in vitro PTC drug sensitivity screenning — The choice of chemotherapy is based on the PTC drug sensitivity results.
  Other Names: docetaxel and trastuzumab and pertuzumab; docetaxel and carboplatin and trastuzumab and pertuzumab

SUMMARY:
Neoadjuvant treatment is an important treatment for early breast cancer patients. Patients with her2 enriched subtype who achieved pCR after neoadjuvant treatment would have longer survival. The neoadjuvant treatment for her2 positive patients include chemotherapy and targeted therapy. Although the pCR rate was high to 60% after use of trastuzumab and pertuzumab, but the adverse reaction of combined chemotherapy could not be negligible. Some studies have attempted chemotherapy-free treatment for her2 positive patients during neoadjuvant therapy. But, which patient could be exempted from chemotherapy and which drug could be omitted are still unknow before treatment. Drug sensitivity screening in vitro was a promising method for choosing chemotherapy. But there was no method could select effective drugs accurately for breast cancer patients until now.

Previously, investigators developed a patient-derived tumor-like cell clusters in vitro culture technology. Feasibility for guiding clinical treatment by drug sensitivity screening based on this technology have been explored by preliminary exploration with a well corresponding. And the results have been published. This study will explore whether drug screening in vitro patient-derived tumor-like cell clusters from breast cancer tissue could be a metheod for omitting chemotherapy for her2 positive participants.

DETAILED DESCRIPTION:
Neoadjuvant chemotherapy for breast cancer could make unresectable breast cancer be resectable and improve breast conservation rate. Patients with her2 enriched subtype who achieved pCR after neoadjuvant treatment would have longer survival. The neoadjuvant treatment for her2 positive patients include chemotherapy and targeted therapy. Although the pCR rate was high to 60% after use of trastuzumab and pertuzumab, but the adverse reaction of combined chemotherapy could not be negligible. Based on the application of dual targeted drugs, some studies have attempted chemotherapy-free treatment for her2 positive patients during neoadjuvant therapy. But, which patient could be exempted from chemotherapy and which drug could be omitted are still unknow before treatment. Drug sensitivity screening in vitro was a promising method for choosing chemotherapy. But there was no method could select effective drugs accurately for breast cancer participants until now.

Previously, investigators developed a patient-derived tumor-like cell clusters(PTC) in vitro culture technology. It is a cell cluster including tumor cells, mesenchymal cells and lymphocytes, which simulates the tumor microenvironment in vitro. In the preliminary exploration, investigators included 35 early breast cancer participants, the corresponding between in vitro drug sensitivity screening based on this technology and clinical treatment results was well. The results have been published.

This study will focus on her2 positive early breast cancer participants. 46 participants will be included. All of them will received in vitro drug sensitivity screenning upon PTC before neoadjuvant therapy. All participants will received trastuzumab and pertuzumab. The choice of chemotherapy drugs is determined based on the PTC drug sensitivity results. If single-agent chemotherapy is effective in vitro, this drug will be the chemotherapy regimen for the corresponding participants. This study expects that the pCR rate could achieve 60% in the case of chemotherapy downgrading after in vitro drug sensitivity screening.

ELIGIBILITY:
Inclusion Criteria:

* invasive breast cancer
* HER2 positive
* T2 or node positive
* ECOG 0-1

Exclusion Criteria:

* stage IV
* inflammatory breast cancer
* Severe chronic disease

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-03-28 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
pathological complete response(pCR) | up to 12 weeks
  ypT0/is, ypN0

SECONDARY OUTCOMES:
event-free survival (EFS) | 5 years
  The time from random assignment to disease progression, including local progression before surgery; disease recurrence-local, regional, distant, ipsilateral noninvasive, or contralateral (invasive or noninvasive)-or death from any cause
invasive disease-free survival(IDFS) | 5 years
  The time from surgery to the first documented occurrence of an event defined as ipsilateral invasive local recurrence, ipsilateral locoregional invasive recurrence, distant recurrence, contralateral invasive breast cancer, or death from any cause
objective response rate | up to 12 weeks
  complete response and partial response

CONTACTS AND LOCATIONS:
Overall Officials: Shu Wang, doctor, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People'S Hospital, Beijing, Beijing Municipality, China